CLINICAL TRIAL: NCT00473187
Title: Effects of Growth Hormone Treatment on Body Proportions and Final Height Among Small Children With X-Linked Hypophosphatemic Rickets
Brief Title: Effects of GH on Body Proportions and Final Height in X-Linked Hypophosphatemic Rickets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rostock (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKJ-Haffner-XLHR-08-2004
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Hypophosphatemic Rickets; Growth Disorders; Somatropin Therapy
Keywords: X-linked dominant hypophosphatemic rickets; growth disorders; anthropometry; human growth hormone
MeSH Terms: conditions — Rickets, Hypophosphatemic; Growth Disorders; Familial Hypophosphatemic Rickets | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: somatropin

SUMMARY:
X-linked hypophosphatemic rickets (XLH) is characterized by rickets, disproportionate short stature, impaired renal phosphate reabsorption and vitamin D metabolism. Despite oral phosphate and vitamin D treatment, most children with XLH demonstrate reduced adult height. The main objective of the study is to determine the beneficial effects of recombinant human growth hormone (rhGH) therapy on body proportions after 36 month in these patients. Secondary objective is to monitor side effects of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Tanner stages of puberty B1, G1
* body height < 2,5 SDS
* growth velocity < 75%
* confirmed diagnosis of XLHR
* conservative treatment for at least 1 year (phosphate, vitamin D)
* informed consent, written agreement

Exclusion Criteria:

* growth hormone deficiency
* hypothyreosis
* severe rickets
* severe physical deformities
* severe hyperparathyreoidism
* chronic renal failure
* complex syndrome involving failure to thrive
* chronic disease with failure to thrive
* impairment of glucose tolerance
* Tanner stages of puberty greater than B1, G1
* medical history of malignancy
* therapy with growth hormone, glucocorticoides, anabolica
* attending another clinical trial

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-08; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
change of body proportion and final height | within 5 years

SECONDARY OUTCOMES:
side effects of therapy with rhGH | within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schnabel, MD, Principal Investigator — University Childrens Hospital - Charite, Berlin; Hagen Staude, Principal Investigator — University Childrens Hospital, Rostock; Dieter Haffner, MD, Principal Investigator — University Childrens Hospital, Rostock
Locations (1):
- University Childrens Hospital, Rostock, Rostock, Mecklenburg-Vorpommern, Germany